CLINICAL TRIAL: NCT04661644
Title: A Phase 1/2a Clinical Trial to Evaluate the Efficacy and Safety of Allogenic Adipose Tissue-derived Mesenchymal Stem Cell Clusters in Patients with Critical Limb Ischemia
Brief Title: Efficacy and Safety of Mesenchymal Stem Cell Clusters in Patients with Critical Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.Biomedics Co., Ltd. (Industry)
Collaborators: Dt&Sanomedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SB-AC-001
Record Dates: First submitted 2020-11-20; First posted 2020-12-10 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Critical Limb Ischemia
Keywords: Adipose-derived mesenchymal stem cells; Critical limb ischemia; Stem cells; Ischemia; S.Biomedics
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Ischemia

STUDY DESIGN:
Intervention Model Description: Phase 1 is conducted to evaluate the tolerability of the IP Subjects receive the IP once and are checked for adverse events. Subjects are evaluated for adverse events after the administration of the IP by registering 3 subjects each at the dosing phase.
  If the maximum tolerated dose (MTD) is determined with the test group 2 (high dose) in the Phase 1, the Phase 2a clinical trial will be conducted. However, if 1 adverse events occur, the test group 2 will be considered as the maximum tolerated dose (MTD), or but only the test group 1 will proceed to Phase 2a.
  If 2 adverse events occur, a dose smaller than test group 1 (low dose) is determined to be the maximum tolerated dose. The Phase 2a clinical trial will not proceed and the clinical trial will end.
  If tolerability and safety are secured, subjects meeting the final inclusion criteria are assigned to Phase 2a, admitted by the same procedure, and administered the IP once. Safety and efficacy assessments are performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group 1 (Low Dose) (Experimental): - Administration Method: 1 mL is withdrawn from 1 vial of clusters of adipose-derived mesenchymal stem cells, composed of adipose-derived mesenchymal stem cells and diluted with 20 mL of saline, which is divided into 1 cc pre-filled syringes and administered in 20 divided doses to 15-20 parts of the muscle in divided doses along the working areacourse of the tibial artery and peroneal artery below the knee joint (above the lower ischemic area) of the subject (above the lower ischemic area) of the subjects under general anesthesia or spinal anesthesia so that the entire diluted solution is administered.
  Interventions: Biological: Clusters of adipose-derived mesenchymal stem cells (Dose: 1 x 10^7 cells/1 mL/vial)
- Test Group 2 (High Dose) (Experimental): - Administration Method: 1 mL is withdrawn from 1 vial of clusters of adipose-derived mesenchymal stem cells, composed of adipose-derived mesenchymal stem cells and diluted with 20 mL of saline, then administered to 15-20 parts of the muscle along the working areacourse of the tibial artery and peroneal artery below the knee joint (above the lower ischemic area) of the subject (above the lower ischemic area) of the subjects under general anesthesia or spinal anesthesia.
  Interventions: Biological: Clusters of adipose-derived mesenchymal stem cells (Dose: 1 x 10^8 cells/1 mL/vial)

INTERVENTIONS:
Biological: Clusters of adipose-derived mesenchymal stem cells (Dose: 1 x 10^7 cells/1 mL/vial) — Dose: 1 x 10^7 cells/1 mL/vial (1,000 clusters of adipose-derived mesenchymal stem cells)
  Arms: Test Group 1 (Low Dose)
Biological: Clusters of adipose-derived mesenchymal stem cells (Dose: 1 x 10^8 cells/1 mL/vial) — Dose: 1 x 10^8 cells/1 mL/vial (10,000 clusters of adipose-derived mesenchymal stem cells)
  Arms: Test Group 2 (High Dose)

SUMMARY:
This clinical trial is designed as a Phase 1/2a clinical trial targeting patients with critical limb ischemia. The trial is composed of Phase 1 to assess the tolerability and safety and Phase 2a to assess the safety and efficacy of the investigational product(A cluster of adipose-derived mesenchymal stem cells (3D-A) (cluster of adipose- derived mesenchymal stem cells)) and proceeds in that order.

DETAILED DESCRIPTION:
This clinical trial is designed as a Phase 1/2a clinical trial targeting patients with critical limb ischemia. The trial is composed of Phase 1 to assess the tolerability and safety and Phase 2a to assess the safety and efficacy of the investigational product.

Phase 1: Open-label, 3 + 3 design, single-center This phase is conducted in a 3 + 3 design by dose level to evaluate the tolerability of the investigational product.

If the subject voluntarily agrees signs the informed consent formin writing to participate in this clinical trial, the subjects who had necessary check-ups and tests and meet the inclusion criteria after subject conformity assessment are registered in the clinical trial.The subjects receive the investigational product once and are checked for adverse events through day 1 and then discharged. The safety and efficacy assessments are conducted through visits at week 4, week 12, and week 24 after administration.

Subjects are evaluated for adverse events up to week 4 after the administration of the investigational product by registering 3 subjects each at the dosing phase. This evaluation is conducted according to the number of persons subjects who developed Grade 3 or higher adverse drug reactions (ADRs) according to CTCAE Version_5.0 in which a causal relation with the investigational product cannot be ruled out.

If the maximum tolerated dose (MTD) is determined with the test group 2 (high dose) in the Phase 1 clinical trial, the Phase 2a clinical trial will be conducted with the two groups, test group 2 and test group 1.

However, if adverse events occur in 1 of 6 subjects, the test group 2 will be decided considered as the maximum tolerated dose (MTD), or but only the test group 1 will proceed to Phase 2a.

If adverse events occur in 2 or more subjects out of 6 subjects, a dose smaller than test group 1 (low dose) is determined to be the maximum tolerated dose. The Phase 2a clinical trial will not proceed and the clinical trial will end.

Phase 2a: Open-label, sequential assignment, single-center If tolerability and safety are secured 4 weeks after administration of the investigational product of Phase 1, Phase 2a is conducted.

Only those subjects meeting the final inclusion criteria are sequentially assigned, admitted by the same procedure, and administered the investigational product once. Subjects are checked for adverse events through day 1 and discharged. Safety and efficacy assessments are performed at week 4, week 12, and week 24 after administration. All subjects are tested with the same schedule, excluding their doses.

The subjects enrolled in Phase 1 are analyzed for efficacy through visits at week 12 and week 24 so that all subjects (Phase 1 and Phase 2a) are assessed and analyzed for efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 or older
2. A person diagnosed with critical limb ischemia due to peripheral artery stenosis or obstructive occlusive disease (Rutherford category 4, 5, 6)
3. Patients with critical limb ischemia where symptoms do not improve even after medication treatment for more than 3 months[1]
4. Persons who voluntarily agreed to participate in this clinical trial

Exclusion Criteria:

1. Persons whose life expectancy is less than 6 months
2. Patients who underwent surgery and interventional procedures (percutaneous vascular intervention, vascular reconstruction, etc.) in the same disease within 3 months of screening
3. Patients in need of interventional procedure or surgery
4. Patients with a history of administration of other cell therapy products
5. Persons who have received systemic immunosuppression treatment within 3 months of screening
6. Persons with a history of a malignant tumor within 5 years of screening (However, non-metastatic basal cell skin carcinoma, squamous cell carcinoma of the skin or carcinoma in situ of the cervix that does not recur for at least 1 year before the registration are excluded)
7. Persons with a hematologic disease with major bleeding or bleeding predisposition within 3 months of screening
8. Women who are pregnant, breastfeeding or planning to become pregnant during the clinical trial period or women of childbearing potential who do not use medically acceptable birth control

   *Medically acceptable contraception:
   * Medicine: Oral contraceptives, skin patches or progestin medications (Transplant or injection)
   * Diaphragm: Condoms, diaphragms, intrauterine devices (IUDs), vaginal suppositories
   * Abstinence: Absolute abstinence (However, periodic abstinence (e.g., calendar method, ovulation method, sympto-thermal method) and control are not considered acceptable contraceptive methods.)
9. Persons who participated in other clinical trials within 3 months of screening
10. Persons who were administered prohibited concomitant medications related to this clinical trial
11. Persons with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels more than twice the normal upper limit at the time of screening
12. Persons identified with estimated glomerular filtration rate (eGFR) levels < 30 mL/min/1.73 m2 at the time of screening
13. Persons with a history of allergies or hypersensitivity to the investigational product or its components
14. Persons who are judged to be inadequate to participate in clinical trials by other investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in ischemic pain | The degrees of changes in VAS measurement on week 4, week 12, week 24, compared to the baseline.
  Changes in 10 cm VAS (Visual analog score) measurement shall be recorded, and statistically analyzed (mean, median, max, min, STD, average). The degree of change shall be compared between the test groups using two sample t-test or Wilcoxon's rank sum test)
Changes in pain-free walking distance | The degrees of changes in pain-free walking distance on week 4, week 12, week 24, compared to the baseline.
  Changes in maximum walking distance on a treadmill shall be measured, and statistically analyzed(mean, median, max, min, STD, average). The degree of change shall be compared between the test groups using two sample t-test or Wilcoxon's rank sum test)
Changes in TBI (Toe Brachial Index) | The degrees of changes in TBI on week 4, week 12, week 24, compared to the baseline.
  Changes in TBI (Toe Brachial Index) shall be recorded, and statistically analyzed (mean, median, max, min, STD, average). The degree of change shall be compared between the test groups using two sample t-test or Wilcoxon's rank sum test)
Changes in ABI (Ankle Brachial Index) | The degrees of changes in ABI on week 4, week 12, week 24, compared to the baseline.
  Changes in ABI (Ankle Brachial Index) shall be recorded, and statistically analyzed (mean, median, max, min, STD, average). The degree of change shall be compared between the test groups using two sample t-test or Wilcoxon's rank sum test)
Change in size of the Ulcer | The degrees of changes in Ulcer size on week 4, week 12, week 24, compared to the baseline.
  The size of the largest ulcer shall be measured and statistically analyzed (mean, median, max, min, STD, average). The degree of change shall be compared between the test groups using two sample t-test or Wilcoxon's rank sum test)
Determination of maximum tolerable dose according to DLT occurrence | Occurrence of ADR is monitored throughout the baseline to week 4 during phase 1.
  Occurrence of adverse drug reactions that are definitely related to the administrated drug are monitored. Maximum tolerable dose is determined when ADR with grade 3 or higher with accordance to CTCAE version 5.0 has occurred to at least one of the three subjects.
Incidence of abnormal laboratory tests results | Laboratory tests are performed on screening(-4~-2 week), baseline, 1 day after the baseline, and on week 4, week 12, week 24, compared to the baseline.
  The following laboratory tests are conducted. In case the results are abnormal, it shall be recorded as a adverse event or excluded from study (screening).
  Hematologic Test: WBC, RBC, Hemoglobin, Hematocrit, Platelets count, Blast, Promyelocyte, Metamyelocyte, Neutrophil (Seg, Band), Eosinophil, Basophil, Lymphocyte, Monocyte, Atypical Lymphocyte, Immature cell, Plasma cell, Nucleated RBC, Abnormal lymphoid cell Blood Chemistry Test: Total protein, Albumin, Globulin, Total Bilirubin, AST, ALT, ALP, BUN, Creatinine, Glucose, Uric Acid, Estimated GFR, Ca, P, CRP, CPK Urine Test: Specific gravity, pH, Glucose, Albumin, Bilirubin, Urobilinogen, Ketone, Blood, Nitrite, Leukocyte Esterase
Incidence of abnormal blood pressure | Blood pressure is measured throughout the study (on screening visit(4~2 week before the baseline), base line, a day after the baseline, week 4, 12, 24 compared to the baseline.)
  Systolic/Diastolic blood pressure is measured after relaxing in sitted position for 5 minutes. In case the results are clinically abnormal, it shall be recorded as an adverse event or excluded from study (screening).
Incidence of abnormal temperature | Temperature is measured throughout the study (on screening visit(4~2 week before the baseline), base line, a day after the baseline, week 4, 12, 24 compared to the baseline.)
  Temperature is measured via eardrum after relaxing in sitted position for 5 minutes. In case the results are clinically abnormal, it shall be recorded as an adverse event.
Incidence of abnormal physical condition | Examined on every visits, throughout the study (on screening visit(4~2 week before the baseline), base line, a day after the baseline, week 4, 12, 24 compared to the baseline.)
  Appearance, skin, head, neck, heart, stomach, urology system, reproductive system, limbs, musculoskeletal system, nervous system, lymphatic glands and etc are examined. In case any clinically abnormal condition has been monitored, it shall be recorded as an adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ik Kim, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isner JM, Baumgartner I, Rauh G, Schainfeld R, Blair R, Manor O, Razvi S, Symes JF. Treatment of thromboangiitis obliterans (Buerger's disease) by intramuscular gene transfer of vascular endothelial growth factor: preliminary clinical results. J Vasc Surg. 1998 Dec;28(6):964-73; discussion 73-5. doi: 10.1016/s0741-5214(98)70022-9. PMID 9845647
- [Background] Bura A, Planat-Benard V, Bourin P, Silvestre JS, Gross F, Grolleau JL, Saint-Lebese B, Peyrafitte JA, Fleury S, Gadelorge M, Taurand M, Dupuis-Coronas S, Leobon B, Casteilla L. Phase I trial: the use of autologous cultured adipose-derived stroma/stem cells to treat patients with non-revascularizable critical limb ischemia. Cytotherapy. 2014 Feb;16(2):245-57. doi: 10.1016/j.jcyt.2013.11.011. PMID 24438903
- [Background] Powell RJ, Goodney P, Mendelsohn FO, Moen EK, Annex BH; HGF-0205 Trial Investigators. Safety and efficacy of patient specific intramuscular injection of HGF plasmid gene therapy on limb perfusion and wound healing in patients with ischemic lower extremity ulceration: results of the HGF-0205 trial. J Vasc Surg. 2010 Dec;52(6):1525-30. doi: 10.1016/j.jvs.2010.07.044. PMID 21146749
- [Background] Lee HC, An SG, Lee HW, Park JS, Cha KS, Hong TJ, Park JH, Lee SY, Kim SP, Kim YD, Chung SW, Bae YC, Shin YB, Kim JI, Jung JS. Safety and effect of adipose tissue-derived stem cell implantation in patients with critical limb ischemia: a pilot study. Circ J. 2012;76(7):1750-60. doi: 10.1253/circj.cj-11-1135. Epub 2012 Apr 12. PMID 22498564
- [Background] Murphy MP, Lawson JH, Rapp BM, Dalsing MC, Klein J, Wilson MG, Hutchins GD, March KL. Autologous bone marrow mononuclear cell therapy is safe and promotes amputation-free survival in patients with critical limb ischemia. J Vasc Surg. 2011 Jun;53(6):1565-74.e1. doi: 10.1016/j.jvs.2011.01.074. Epub 2011 Apr 22. PMID 21514773
- [Background] Lasala GP, Silva JA, Minguell JJ. Therapeutic angiogenesis in patients with severe limb ischemia by transplantation of a combination stem cell product. J Thorac Cardiovasc Surg. 2012 Aug;144(2):377-82. doi: 10.1016/j.jtcvs.2011.08.053. Epub 2011 Nov 12. PMID 22079876
- [Background] Kawamoto A, Katayama M, Handa N, Kinoshita M, Takano H, Horii M, Sadamoto K, Yokoyama A, Yamanaka T, Onodera R, Kuroda A, Baba R, Kaneko Y, Tsukie T, Kurimoto Y, Okada Y, Kihara Y, Morioka S, Fukushima M, Asahara T. Intramuscular transplantation of G-CSF-mobilized CD34(+) cells in patients with critical limb ischemia: a phase I/IIa, multicenter, single-blinded, dose-escalation clinical trial. Stem Cells. 2009 Nov;27(11):2857-64. doi: 10.1002/stem.207. PMID 19711453
- [Background] Ruiz-Salmeron R, de la Cuesta-Diaz A, Constantino-Bermejo M, Perez-Camacho I, Marcos-Sanchez F, Hmadcha A, Soria B. Angiographic demonstration of neoangiogenesis after intra-arterial infusion of autologous bone marrow mononuclear cells in diabetic patients with critical limb ischemia. Cell Transplant. 2011;20(10):1629-39. doi: 10.3727/096368910X0177. PMID 22289660
- [Background] Benoit E, O'Donnell TF, Patel AN. Safety and efficacy of autologous cell therapy in critical limb ischemia: a systematic review. Cell Transplant. 2013;22(3):545-62. doi: 10.3727/096368912X636777. Epub 2012 Mar 28. PMID 22490340
- [Background] Cacione DG, do Carmo Novaes F, Moreno DH. Stem cell therapy for treatment of thromboangiitis obliterans (Buerger's disease). Cochrane Database Syst Rev. 2018 Oct 31;10(10):CD012794. doi: 10.1002/14651858.CD012794.pub2. PMID 30378681
- [Background] Criqui MH, Fronek A, Barrett-Connor E, Klauber MR, Gabriel S, Goodman D. The prevalence of peripheral arterial disease in a defined population. Circulation. 1985 Mar;71(3):510-5. doi: 10.1161/01.cir.71.3.510. PMID 3156006
- [Background] Selvin E, Erlinger TP. Prevalence of and risk factors for peripheral arterial disease in the United States: results from the National Health and Nutrition Examination Survey, 1999-2000. Circulation. 2004 Aug 10;110(6):738-43. doi: 10.1161/01.CIR.0000137913.26087.F0. Epub 2004 Jul 19. PMID 15262830
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Kinlay S. Management of Critical Limb Ischemia. Circ Cardiovasc Interv. 2016 Feb;9(2):e001946. doi: 10.1161/CIRCINTERVENTIONS.115.001946. PMID 26858079
- [Background] Dohmen A, Eder S, Euringer W, Zeller T, Beyersdorf F. Chronic critical limb ischemia. Dtsch Arztebl Int. 2012 Feb;109(6):95-101. doi: 10.3238/arztebl.2012.0095. Epub 2012 Feb 10. PMID 22396707
- [Background] Davies MG. Criticial limb ischemia: epidemiology. Methodist Debakey Cardiovasc J. 2012 Oct-Dec;8(4):10-4. doi: 10.14797/mdcj-8-4-10. PMID 23342182
- [Background] Soder HK, Manninen HI, Jaakkola P, Matsi PJ, Rasanen HT, Kaukanen E, Loponen P, Soimakallio S. Prospective trial of infrapopliteal artery balloon angioplasty for critical limb ischemia: angiographic and clinical results. J Vasc Interv Radiol. 2000 Sep;11(8):1021-31. doi: 10.1016/s1051-0443(07)61332-3. PMID 10997465
- [Background] Nasr MK, McCarthy RJ, Hardman J, Chalmers A, Horrocks M. The increasing role of percutaneous transluminal angioplasty in the primary management of critical limb ischaemia. Eur J Vasc Endovasc Surg. 2002 May;23(5):398-403. doi: 10.1053/ejvs.2002.1615. PMID 12027466
- [Background] Guiducci S, Porta F, Saccardi R, Guidi S, Ibba-Manneschi L, Manetti M, Mazzanti B, Dal Pozzo S, Milia AF, Bellando-Randone S, Miniati I, Fiori G, Fontana R, Amanzi L, Braschi F, Bosi A, Matucci-Cerinic M. Autologous mesenchymal stem cells foster revascularization of ischemic limbs in systemic sclerosis: a case report. Ann Intern Med. 2010 Nov 16;153(10):650-4. doi: 10.7326/0003-4819-153-10-201011160-00007. PMID 21079220
- [Background] Gupta PK, Chullikana A, Parakh R, Desai S, Das A, Gottipamula S, Krishnamurthy S, Anthony N, Pherwani A, Majumdar AS. A double blind randomized placebo controlled phase I/II study assessing the safety and efficacy of allogeneic bone marrow derived mesenchymal stem cell in critical limb ischemia. J Transl Med. 2013 Jun 10;11:143. doi: 10.1186/1479-5876-11-143. PMID 23758736
- [Background] Ito J, Moriyama H, Inokuchi S, Goto N. Human lower limb muscles: an evaluation of weight and fiber size. Okajimas Folia Anat Jpn. 2003 Aug;80(2-3):47-55. doi: 10.2535/ofaj.80.47. PMID 14604153
- [Background] Charles JP, Cappellari O, Spence AJ, Hutchinson JR, Wells DJ. Musculoskeletal Geometry, Muscle Architecture and Functional Specialisations of the Mouse Hindlimb. PLoS One. 2016 Apr 26;11(4):e0147669. doi: 10.1371/journal.pone.0147669. eCollection 2016. PMID 27115354
- [Background] Park IS, Rhie JW, Kim SH. A novel three-dimensional adipose-derived stem cell cluster for vascular regeneration in ischemic tissue. Cytotherapy. 2014 Apr;16(4):508-22. doi: 10.1016/j.jcyt.2013.08.011. Epub 2013 Nov 7. PMID 24210783
- [Background] Park IS, Kang JA, Kang J, Rhie JW, Kim SH. Therapeutic effect of human adipose-derived stromal cells cluster in rat hind-limb ischemia. Anat Rec (Hoboken). 2014 Dec;297(12):2289-98. doi: 10.1002/ar.22961. Epub 2014 Jul 25. PMID 25066828
- [Background] Schroder F, Diehm N, Kareem S, Ames M, Pira A, Zwettler U, Lawall H, Diehm C. A modified calculation of ankle-brachial pressure index is far more sensitive in the detection of peripheral arterial disease. J Vasc Surg. 2006 Sep;44(3):531-6. doi: 10.1016/j.jvs.2006.05.016. PMID 16950430
- [Background] Rutherford RB, Baker JD, Ernst C, Johnston KW, Porter JM, Ahn S, Jones DN. Recommended standards for reports dealing with lower extremity ischemia: revised version. J Vasc Surg. 1997 Sep;26(3):517-38. doi: 10.1016/s0741-5214(97)70045-4. PMID 9308598
- [Background] Heo SH, Park YS, Kang ES, Park KB, Do YS, Kang KS, Kim DI. Early Results of Clinical Application of Autologous Whole Bone Marrow Stem Cell Transplantation for Critical Limb Ischemia with Buerger's Disease. Sci Rep. 2016 Jan 21;6:19690. doi: 10.1038/srep19690. PMID 26791280
- [Background] Kim HJ, Jang SY, Park JI, Byun J, Kim DI, Do YS, Kim JM, Kim S, Kim BM, Kim WB, Kim DK. Vascular endothelial growth factor-induced angiogenic gene therapy in patients with peripheral artery disease. Exp Mol Med. 2004 Aug 31;36(4):336-44. doi: 10.1038/emm.2004.44. PMID 15365252
- [Background] Qadura M, Terenzi DC, Verma S, Al-Omran M, Hess DA. Concise Review: Cell Therapy for Critical Limb Ischemia: An Integrated Review of Preclinical and Clinical Studies. Stem Cells. 2018 Feb;36(2):161-171. doi: 10.1002/stem.2751. Epub 2018 Jan 3. PMID 29226477
- [Background] Greenblatt DJ, Allen MD. Intramuscular injection-site complications. JAMA. 1978 Aug 11;240(6):542-4. PMID 671665
- [Background] Muller-Vahl H. Adverse reactions after intramuscular injections. Lancet. 1983 May 7;1(8332):1050. doi: 10.1016/s0140-6736(83)92679-x. No abstract available. PMID 6133092
- [Background] Mishra P, Stringer MD. Sciatic nerve injury from intramuscular injection: a persistent and global problem. Int J Clin Pract. 2010 Oct;64(11):1573-1579. doi: 10.1111/j.1742-1241.2009.02177.x. PMID 20670272
- [Background] Rodger MA, King L. Drawing up and administering intramuscular injections: a review of the literature. J Adv Nurs. 2000 Mar;31(3):574-82. doi: 10.1046/j.1365-2648.2000.01312.x. PMID 10718876
- [Background] Cocoman A, Murray J. Intramuscular injections: a review of best practice for mental health nurses. J Psychiatr Ment Health Nurs. 2008 Jun;15(5):424-34. doi: 10.1111/j.1365-2850.2007.01236.x. PMID 18454829
- [Background] Grenon SM, Vittinghoff E, Owens CD, Conte MS, Whooley M, Cohen BE. Peripheral artery disease and risk of cardiovascular events in patients with coronary artery disease: insights from the Heart and Soul Study. Vasc Med. 2013 Aug;18(4):176-84. doi: 10.1177/1358863X13493825. Epub 2013 Jul 8. PMID 23835937
- [Background] Conte MS, Geraghty PJ, Bradbury AW, Hevelone ND, Lipsitz SR, Moneta GL, Nehler MR, Powell RJ, Sidawy AN. Suggested objective performance goals and clinical trial design for evaluating catheter-based treatment of critical limb ischemia. J Vasc Surg. 2009 Dec;50(6):1462-73.e1-3. doi: 10.1016/j.jvs.2009.09.044. Epub 2009 Nov 7. PMID 19897335
- [Background] Shigematsu H, Yasuda K, Iwai T, Sasajima T, Ishimaru S, Ohashi Y, Yamaguchi T, Ogihara T, Morishita R. Randomized, double-blind, placebo-controlled clinical trial of hepatocyte growth factor plasmid for critical limb ischemia. Gene Ther. 2010 Sep;17(9):1152-61. doi: 10.1038/gt.2010.51. Epub 2010 Apr 15. PMID 20393508
- [Derived] Dubsky M, Husakova J, Sojakova D, Fejfarova V, Jude EB. Cell Therapy of Severe Ischemia in People with Diabetic Foot Ulcers-Do We Have Enough Evidence? Mol Diagn Ther. 2023 Nov;27(6):673-683. doi: 10.1007/s40291-023-00667-w. Epub 2023 Sep 22. PMID 37740111